CLINICAL TRIAL: NCT06196983
Title: Effects of Rhythmic Aerobic Exercises on Functional Balance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0731
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group, Rhythmic aerobic exercises (Experimental): Rhythmic aerobic exercises were used in experimental group.
  Interventions: Other: Rhythmic aerobic exercises
- control group, strength and balance exercises (Active Comparator): only strength and balance exercises were given to control group.
  Interventions: Other: Control group, strength and balance exercises

INTERVENTIONS:
Other: Rhythmic aerobic exercises — The experimental group's pattern of functional movements includes both right and left foot movements. To improve muscle strength and the capacity to maintain balance, exercises including running in place, side steps, walking while eating, and turning in place can also be used. The rhythmic aerobic group linked their motions to the rhythmic auditory stimuli in order to perform in a rhythmic manner.
  Arms: Experimental group, Rhythmic aerobic exercises
Other: Control group, strength and balance exercises — The control group engaged in strength and balance exercises where they stood with weight on one leg and raised the other leg to the side or back. In a tandem stance, place your foot heel directly in front of your toe. Get out of a chair, then take a seat without using your hands.
  Arms: control group, strength and balance exercises

SUMMARY:
Down syndrome (DS) is the most commonly occurring chromosomal condition and it affects more than 400,000 people in the United States. The chances of having a child with DS increases as the mother ages. DS is a chromosomal disorder characterized by trisomy 21. These alterations are responsible for motor and cognitive development delay, due to abnormalities on the maturation of the central nervous system. DS presents generalized muscle hypotonia which interferes in motor coordination and postural reactions leading to changes in balance. Rhythmic aerobic exercises for people with intellectual disability are helpful. In these exercises body's large muscles move in a rhythmic manner for a sustained period of time. The aim of this study is to determine the effect of rhythmic aerobic exercises for improving functional balance in children with DS.

This will be a randomized controlled trial study. Study will be approved by ethical committee. After that informed consent will be taken and patients will be included in the study based on the inclusion criteria. 40 patients will be divided into two groups, interventions will be performed for 50 minutes per session twice a week for total of 8 weeks; In experimental group, rhythmic aerobic exercises will be performed. The rhythmic training group initially used rhythmic auditory stimulation with 8 beats, then progressed to 16 beats per minutes. In control group, strength and balance exercises will be performed. Functional balance of the patient will be assessed by checking the quality of Sit-to-stand and Stand to-Sit on the respective sections of Pediatric Balance Scale and Time Up and Go test. Data will be analyzed using SPSS 25. Mean and standard deviation will be calculated. Both groups will be compared by appropriate test.

DETAILED DESCRIPTION:
This will be a randomized controlled trial study. Study will be approved by ethical committee. After that informed consent will be taken and patients will be included in the study based on the inclusion criteria. 40 patients will be divided into two groups, interventions will be performed for 50 minutes per session twice a week for total of 8 weeks; In experimental group, rhythmic aerobic exercises will be performed. The rhythmic training group initially used rhythmic auditory stimulation with 8 beats, then progressed to 16 beats per minutes. In control group, strength and balance exercises will be performed. Functional balance of the patient will be assessed by checking the quality of Sit-to-stand and Stand to-Sit on the respective sections of Pediatric Balance Scale and Time Up and Go test. Data will be analyzed using SPSS 25. Mean and standard deviation will be calculated. Both groups will be compared by appropriate test.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome children
* Aged 9- to 14-year-old
* Functional ability sufficient to understand conversation, exercise guidance and direction
* Have ability to walk 60 meters independently according to 6 minute walk test

Exclusion Criteria:

* Patients did not adapt to the training program, or were not willing to participate in the study
* Did not have ability to stand and walk independently
* Did not have ability to follow simple verbal instructions
* Participants with intellectual disabilities, such as those caused by encephalitis, meningitis, disorders due to metabolic disorders, vitamin deficiency, and tumors were excluded from the study

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pediatric balance scale (PBS) | 8 weeks
  Pediatric balance scale is a modified version of berg balance scale that is used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Time up and go test (TUG) | 8 weeks
  The TUG test measure is the time taken, in seconds, by an individual to stand up from a standard arm chair, walk a distance of 3 m, turn, walk back to the chair, and sit down again.

CONTACTS AND LOCATIONS:
Overall Officials: Laraib -un-Nisa, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vazou S, Klesel B, Lakes KD, Smiley A. Rhythmic Physical Activity Intervention: Exploring Feasibility and Effectiveness in Improving Motor and Executive Function Skills in Children. Front Psychol. 2020 Sep 18;11:556249. doi: 10.3389/fpsyg.2020.556249. eCollection 2020. PMID 33071879
- See also: Rhythmic Physical Activity Intervention: Exploring Feasibility and Effectiveness in Improving Motor and Executive Function Skills in Children. — https://pubmed.ncbi.nlm.nih.gov/33071879/